CLINICAL TRIAL: NCT02976844
Title: Effect of Positive End-expiratory Pressure on Optimal Balloon Volume During Esophageal Pressure Monitoring in Mechanical Ventilated Patients: A Clinical Feasibility Study
Brief Title: Effect of Positive End-expiratory Pressure on Optimal Balloon Volume During Esophageal Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY-2016-11-22
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-01

CONDITIONS: Mechanical Ventilation
Keywords: optimal balloon volume; positive end-expiratory pressure
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low PEEP group: The positive end-expiratory pressure was less than 10cmH2O
  Interventions: Procedure: Positive end-expiratory Pressure
- High PEEP group: The positive end-expiratory pressure was higher or equal to 10cmH2O.
  Interventions: Procedure: Positive end-expiratory Pressure

INTERVENTIONS:
Procedure: Positive end-expiratory Pressure — Positive end-expiratory pressure will be used during mechanical ventilation.

SUMMARY:
Esophageal pressure (PES), which has been used as a surrogate for pleural pressure. The volume of esophageal balloon can influence the accuracy of monitoring esophageal pressure. The optimal balloon volume is directly dependent on surrounding pressure. In the present study,the investigators will observe the optimal volume of esophageal balloon during the different PEEP in bench and clinical study.

DETAILED DESCRIPTION:
The esophageal pressure (Pes) is used as a surrogate for pleural pressure to obtain transpulmonary pressure. Catheter with air balloon is the most commonly used method to measure the Pes. The optimal injected volume of the balloon is the key factor in accurate measurement of Pes. The recoil pressure of the balloon turns up while the balloon is over-filled, resulting in over-estimation of the PES; on the other hand, an under-filled balloon also cannot properly transmit the surrounding pressure of balloon. However, the researchers showed the optimal balloon volumes is related to the surrounding pressure and even is not correspond with manufacturer's recommendations. Theoretically, when balloon transmural pressure(PTM) is zero, representing the balloon in a condition with equivalent pressure inside and outside of the balloon, it was defined as optimal volume. However, in clinical settings, it is difficult to determine the balloon PTM, and therefore the optimal volume cannot be obtained, because the surrounding pressure of the balloon cannot be conveniently measured.

In the present study, the investigators will develop a simple method to obtain the optimal balloon volume and observe the effect of positive end-expiratory pressure on optimal balloon volume during esophageal pressure monitoring. The investigators want to validate the accuracy of method in the bench study and clinical feasibility in mechanical ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* postoperative patients with delayed emergence from general anesthesia admitted to the ICU for mechanical ventilation.

Exclusion Criteria:

* age under 18 years;
* diagnosed or suspected esophageal varices;
* history of chronic obstructive pulmonary diseases or asthma;
* history of esophageal, gastric or lung surgery;
* evidence of active air leak from the lung, including bronchopleural fistula, pneumothorax, pneumomediastinum, or an existing chest tube;
* evidence of severe coagulopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: postoperative patients receiving mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The optimal balloon volume at different PEEP | within 3 minutes after esophageal balloon volume changing
  The 3 minutes after esophageal balloon volume changing, the investigators will record the end-expiratory and end-inspiratory esophageal pressure. The pressure and volume curve will be drawn to determine the optimal volume.

SECONDARY OUTCOMES:
The transpulmonary pressure | within 3 minutes after esophageal balloon volume changing

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sun XM, Chen GQ, Huang HW, He X, Yang YL, Shi ZH, Xu M, Zhou JX. Use of esophageal balloon pressure-volume curve analysis to determine esophageal wall elastance and calibrate raw esophageal pressure: a bench experiment and clinical study. BMC Anesthesiol. 2018 Feb 14;18(1):21. doi: 10.1186/s12871-018-0488-6. PMID 29444644